CLINICAL TRIAL: NCT05943470
Title: The Difference Between Daily and Alternative Day Use of Icodextrin in Peritoneal Dialysis
Brief Title: The Difference Between Daily and Alternative Day Use of Icodextrin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zanzhe Yu, Principal investigator, RenJi Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-083
Record Dates: First submitted 2023-06-11; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Peritoneal Dialysis Solution Adverse Reaction
MeSH Terms: interventions — Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- daily (Active Comparator): daily use of one exchange of icodextin as long dwell
  Interventions: Drug: Icodextrin Peritoneal Dialysis Solution
- alternative day (Experimental): alternative day use of one exchange of icodextin as long dwell
  Interventions: Drug: Icodextrin Peritoneal Dialysis Solution

INTERVENTIONS:
Drug: Icodextrin Peritoneal Dialysis Solution — alternative day use of icodextrin comparing with daily use of icodextrin
  Other Names: Extraneal

SUMMARY:
Volume overload is an important cause of technical failure in peritoneal dialysis patients. Icodextrin can provide continuous ultrafiltration, which provides a new option for peritoneal dialysis patients.

However, icodextrin metabolites are known to accumulate to some extent in the body, resulting in less ultrafiltration with long-term icodextrin use comparing with newly use.

Therefore, the investigator hypothesized that a single dose of icodextrin would produce more ultrafiltration volume with the use of icodextrin dialysate on alternate days than with the use of icodextrin dialysate on daily uses.

DETAILED DESCRIPTION:
1. Patients who met the inclusion criteria will be enrolled in this study.
2. Randomization.
3. Treatment A: daily icodextrin for 2 weeks. Treatment B: icodextrin is used every other day and original glucose-based dialysate is used every other day for a total of 2 weeks. The duration of icodextrin exchange is unchanged from the participants' original dialysate exchange regimen (typically, 8 to 14 hours). The interval is two weeks (the original dialysate was resumed). Participants would receive treatment A-B or B-A, depending on randomization.
4. Participants would record daily peritoneal ultrafiltration volume, long dwell ultrafiltration volume, dialysis prescription, urine volume, body weight, home blood pressure monitoring and complaints of discomfort.
5. Before the start of treatment (day 0), after the end of treatment period 1 (day14), at the end of washout period (day28), and at the end of treatment period 2 (day42), blood samples are collected for blood glucose, blood lipids, BNP, amylase, blood electrolytes, alkaline phosphatase. The participants' weight, blood pressure, dialysis prescription, daily ultrafiltration volume, urine volume, long dwell ultrafiltration volume and BCM measurement results would be recorded on the visit day. In the last 10 enrolled patients, blood samples would be collected for detection of icodextrin metabolites. After the end of treatment period 2, participants could choose the prescription of dialysate according to their own wishes and would be followed up for another 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. End-stage renal failure

  2. Patients with regular peritoneal dialysis in our center

  3. 18-75 years old

  4. Patients who currently use glucose dialysate for prolonged abdominals

  5. Sign informed consent

Exclusion Criteria:

* 1. The expected survival time is less than 3 months

  2. Known peritoneal dialysis tube dysfunction

  3. Peritonitis occurred within one month

  4. Known peritoneal effusion

  5. Known allergy to icodextrin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
ultrafiltration measured in ml | 2 weeks
  ultrafiltration volume for single icodextrin dwell

SECONDARY OUTCOMES:
daily treatment cost measured in Chinese Yuan | 2 weeks
  daily treatment cost

IPD SHARING:
Plan to Share IPD: No